CLINICAL TRIAL: NCT07032441
Title: Association Between Sleep Deprivation and Malnutrition in Intensive Care Unit Patients: A Prospective Observational Cohort Study
Brief Title: Impact of Sleep Deprivation on Malnutrition in ICU (Intensive Care Unit) Patients
Status: Not yet recruiting | Type: Observational
Sponsor: Shanghai Zhongshan Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: SD-ICU-Malnutrition
Record Dates: First submitted 2025-06-11; First posted 2025-06-24 (Actual); Last update posted 2025-06-24 (Actual); Status verified 2025-06

CONDITIONS: ICU Hospitalization; Sleep Deprivation; Malnutrition Severe
MeSH Terms: conditions — Sleep Deprivation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- SD-ICU
  Interventions: Device: PSG

INTERVENTIONS:
Device: PSG — Polysomnography (PSG) is a comprehensive test used to assess sleep disorders and monitor sleep quality. PSG is typically conducted in specialized sleep laboratories and can simultaneously record various physiological parameters to help doctors diagnose different types of sleep disorders, such as obstructive sleep apnea, insomnia, and periodic limb movement disorder.
  The monitored components of PSG usually include:
  Electroencephalogram (EEG): Records the electrical activity of the brain to determine different sleep stages.
  Electrooculogram (EOG): Records eye movements to identify rapid eye movement (REM) sleep stages.
  Electromyogram (EMG): Records muscle activity, typically monitoring the muscles of the jaw or legs.
  Electrocardiogram (ECG): Monitors the electrical activity of the heart. Respiratory flow monitoring: Records the flow and frequency of breathing. Oxygen saturation monitoring: Monitors blood oxygen levels using a pulse oximeter.

SUMMARY:
Study Design This study is a prospective cohort design conducted at Zhongshan Hospital affiliated with Fudan University. It will involve systematic assessments of sleep quality, nutritional status, and associated clinical outcomes in adult ICU patients over a defined observation period.

Sample Size: An estimated 150 adult patients (≥18 years) will be recruited from the ICU.

Assessments 1. Sleep Quality Assessment:

1. Polysomnography (PSG): Sleep quality and duration will be quantified using PSG, which records brain waves, blood oxygen levels, heart rate, and breathing, as well as eye and leg movements. This will provide a comprehensive picture of sleep architecture and disturbances.
2. Sleep Quality Index: In addition to PSG data, the Pittsburgh Sleep Quality Index (PSQI) will be administered to assess subjective sleep quality, sleep latency, duration, habitual sleep efficiency, sleep disturbances, and daytime dysfunction.

2. Nutritional Status Evaluation:

1. Nutritional Risk Screening Tools: The Nutritional Risk Screening (NRS-2002) and the Malnutrition Universal Screening Tool (MUST) will be applied to assess nutritional risk and identify malnutrition.
2. Biochemical Assessment: Blood samples will be collected to measure biochemical indicators such as serum albumin, transferrin, prealbumin, and other relevant markers of nutritional status.
3. Anthropometric Measurements: Body mass index (BMI) and muscle mass assessments will be conducted using bioelectrical impedance analysis (BIA) or dual-energy X-ray absorptiometry (DEXA) to quantify body composition.

3. Physiological Monitoring:

1. Continuous monitoring of vital signs, including heart rate, blood pressure, and respiratory rate, will be performed.
2. Assessment of immune function through laboratory tests, including white blood cell count and levels of inflammatory markers (C-reactive protein).

4. Complications Tracking:

1. Data on complications such as infections, delayed wound healing, and respiratory failure will be systematically recorded throughout the ICU stay.

This study aims to elucidate the complex interplay between sleep deprivation and malnutrition in ICU patients. By identifying key associations and influencing factors, we hope to inform targeted clinical interventions that can improve patient care, recovery, and quality of life. The findings will serve as a foundation for future research exploring the intricate relationships between sleep and nutritional status in critical care settings.

ELIGIBILITY:
Inclusion Criteria:

* Adult ICU patients (≥18 years)
* Expected length of stay ≥5 days
* No severe liver or kidney failure (to avoid confounding in nutritional metabolism)

Exclusion Criteria:

* Pre-existing malnutrition upon admission (e.g., BMI <18.5 or weight loss >10% within 6 months)
* Neuromuscular diseases affecting metabolic assessment

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who met the inclusion criteria in the ICU of Zhongshan Hospital, Fudan University from August 2025 were enrolled.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2025-08-01 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-12-31 (Estimated)

PRIMARY OUTCOMES:
Prevalence of malnutrition | From enrollment to the end of treatment at 8 weeks
  NRS-2002
Changes in physiological indicator | From enrollment to the end of treatment at 8 weeks
  Muscle mass

SECONDARY OUTCOMES:
The length of stay (LOS) in ICU | From enrollment to the end of treatment at 8 weeks
  LOS in ICU is a critical metric in healthcare that reflects the duration a patient spends receiving specialized care in an ICU setting.
Incidence of complications | From enrollment to the end of treatment at 8 weeks
  In ICUs, monitoring the incidence of complications is crucial for assessing patient safety, treatment efficacy, and overall healthcare quality.

IPD SHARING:
Plan to Share IPD: No